CLINICAL TRIAL: NCT03980119
Title: Utilizing the HITSystem 3.0 for Optimizing Paediatric ART Retention and Adherence in Western Nyanza Province, Kenya
Brief Title: Utilizing the HITSystem for Optimizing Paediatric ART Retention and Adherence in Western Nyanza Province, Kenya
Acronym: PARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Global Health Innovations (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HITSystem Peds Retention Kenya
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Pediatric HIV Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HITSystem 3.0 Intervention (Experimental): All HIV-positive children and their caregivers attending health facilities randomized to the HITSystem intervention arm will be monitored by the HITSystem. In the event that the child misses an appointment or a scheduled laboratory test, or the child's laboratory results suggest ART treatment failure, an automated SMS text message and alert will be generated in the HITSystem that will notify the child's health care provider. The child's caregiver will also receive a text message asking them to return to the clinic with the child. If the child is 16 years of age and considered an independent adolescent without a caregiver, the same process will be implemented, with the text messages being sent directly to the child. If the child's caregiver, or the independent adolescent, does not have a mobile phone, the health care provider will notify the community health worker (CHW) to trace the individual and visit them in their home.
  Interventions: Other: HITSystem 3.0
- Control (No Intervention): All HIV-positive children and their caregivers attending health facilities randomized to the Control arm will receive HIV/AIDS standard of care.

INTERVENTIONS:
Other: HITSystem 3.0 — The HITSystem 3.0 is a web-based intervention that aims to improve pediatric ART retention and adherence, and viral suppression. The HITSystem 3.0 is accessed online through a computer, using mobile broadband modems that respond to a cellular signal. The primary components include: (1) action alerts to complete time-sensitive interventions; (2) real time communication of HIV PCR results to hospitals to reduce turn-around time; (3) continuous follow-up for timely ART initiation among HIV-infected infants; (4) promotion of retention in EID care via SMS text messaging and/or patient tracing; and (5) an automated and individualized SMS text messaging component to communicate with mothers. The HITSystem has a unique dashboard that proactively monitors time-sensitive interventions along the EID cascade of care, alerting clinics, laboratories and mothers when an intervention has been missed.
  Arms: HITSystem 3.0 Intervention

SUMMARY:
Overall, there are an estimated 98,000 children living with HIV in Kenya. Children who are initiated on ART in Kenya and other low resource settings face several challenges with ongoing care due to current limitations of paediatric HIV treatment services. High quality paediatric HIV care requires routine monitoring of clinical and virologic status, support for ART adherence, and patient outreach to optimize retention in care.

The HIV Infant Tracking System (HITSystem) is a web-based, system-level intervention that has dramatically improved EID HIV-related outcomes in Kenya, Tanzania, and Malawi.

The objective of this study is to implement and evaluate the impact of HITSystem 3.0 on paediatric clinical outcomes, adherence, retention and viral suppression over 12 months among children in HIV care. Outcome measurements will be evaluated separately in children aged ≤2 years and in those aged 3-16 years.

Primary Outcomes

1. The proportion of HIV infected children in each arm who are retained in HIV care at 12 months. Retention will be defined as regular engagement with HIV care, as measured by having attended the last three scheduled monthly appointments on time (see section 3.3 for further description).
2. The proportion of HIV infected children who are virally suppressed (VL <50) at the end of the 12-month follow-up period.

The proposed trial design is an unblinded CRT with two arms: the HITSystem 3.0 Intervention vs. Standard of Care (SOC) as the control. The CRT will be implemented in 20 health facilities (10 intervention and 10 control) in Western Nyanza province in Kenya and will collect data from HIV-infected children aged ≤16 years. Outcomes will focus on ART retention, adherence and viral suppression.

Outcomes will be assessed among all HIV positive children aged ≤16 years attending the trial facilities for HIV care at the start of the trial, or who are diagnosed as HIV positive during the first 12 months of the trial. Follow-up data will be collected on each child for 12 months. Therefore, the total duration of the trial will be for 24 months.

All HIV-positive children and their caregivers attending health facilities randomised to the intervention arm will be monitored by the HITSystem 3.0.

The study will be conducted in Western Nyanza province, Kenya, which comprises six counties.

ELIGIBILITY:
Inclusion Criteria:

Health facilities must meet the following criteria to be eligible for the trial:

1. Level 3-5 and located in the Western Nyanza Province.
2. Currently provide PMTCT, EID and paediatric ART programmes.
3. Either government or private not-for-profit
4. Agreement to participate, which will be granted by both Kisumu County minister of health, as well as the facility Director of Medical Operations (DMO).

Exclusion Criteria:

1. Facilities that are classified as Level 1-2.
2. Facilities that are participating in other research involving paediatric ART programmes.
3. Private commercial facilities

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1160 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pediatric ART Retention | 12 months
  The proportion of HIV infected children in each arm who are retained in HIV care at 12 months. Retention will be defined as regular engagement with HIV care, as measured by having attended the last three scheduled monthly appointments on time.
Pediatric Viral Load Suppression | 12 months
  The proportion of HIV infected children who are virally suppressed (VL <50) at the end of the 12-month follow-up period.

SECONDARY OUTCOMES:
Missed ART | 12 months
  The proportion of HIV infected children who ever experienced a gap of >30 days without ART medication during the 12-month follow-up period.
Medication Ratio >90% | 12 months
  The proportion of HIV-infected children with an ART medication possession ratio of ≥90% during the 12-month follow-up period
Viral Load Testing | Baseline, 6 months, 12 months
  he proportion of HIV infected children who received viral load testing (per Kenya guidelines) at baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brad Gautney, MPH, Principal Investigator — London School of Hygiene and Tropical Medicine

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available upon publication of results.
Access Criteria: Only PI, appropriate research members and publication editor will have access.